CLINICAL TRIAL: NCT06058858
Title: Incidence and Risks Factors of CMV Reactivation in Patients Receiving of CAR-T Cells for Acute Leukemia and Lymphoma Relapse, a Cohort Study Analysis
Acronym: CMV CAR-T
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APH211589
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Cytomegalovirus Infections; Acute Leukemia; B Cell Lymphoma
MeSH Terms: conditions — Cytomegalovirus Infections; Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Letermovir is approved for the primary prevention of Cytomegalovirus (CMV) reactivation and infection in hematopoietic stem cell transplant recipients. Letermovir may be beneficial in other clinical presentation where CMV reactivates and may alter clinical outcomes. Recently Chimeric Antigen Receptor (CAR) T cells have been used for the treatment of refractory acute leukemia and B cell lymphoma. Reactivation of chronic viral infections, in particular those belonging to the Herpesviridae family can therefore be observed following CAR-T cells treatment.According to first reports, Cytomegalovirus seems to be the main virus detected. Uncontrolled CMV reactivation leads to CMV disease requiring the use of antiviral drugs associated with either hematological toxicity (ganciclovir) or renal toxicity (foscarnet) and is usually associated with poor outcomes. In addition, CMV interplays with the immune system and decreases the immunosurveillance of tumor cells and facilitates the growth or reactivation of other opportunistic infections. Therefore, CMV reactivation could also impact the outcome of CART cells treatment by increasing the existing risk of opportunistic infections in CART cells recipients and thus by increasing morbidity, length stay or require intensive care. Imbalance of the immune system usually correlates with reactivation of persistent virus like Torquetenovirus (TTV), redondovirus or pegivirus found more frequently in Hematopoietic stem-cell transplantation (HSCT) patients or patients requiring intensive care. Whether reactivations of those persistent viruses are associated or precede CMV reactivation deserve careful investigation to identify as early as possible patients at high risk and who could benefit from antiviral preventive treatment.

The objective of this trial is to determine the incidence of CMV reactivation within 3 months after infusion of CAR-T cells in CMV seropositive patients with refractory acute leukemia or B-cell lymphoma.

ELIGIBILITY:
Common inclusion criteria :

* Paediatric (1 to 18 years old) receiving CART-T cells treatment for refractory acute leukemia or B-cell lymphoma
* Adult receiving CART-T cells treatment for refractory acute leukemia or B-cell lymphoma
* CMV seropositive patients

Inclusion criteria : retrospective part

* Provide written non-opposition from the patient signed by investigator
* If the patient is a minor, provide written non-opposition from both parents and child (if age appropriate to collect their non-objection) or child and the legal representative in case only one parent is alive, signed by investigator

Inclusion criteria : prospective part

* Provide written consent form signed by patient and investigator
* If the patient is a minor, provide written consent form signed by investigator and both parents or signed by investigator and the legal representative in case only one parent is alive

Exclusion Criteria:

* CMV seronegative patients
* Lack of affiliation to a social security scheme (as a beneficiary or assignee)
* Patients under guardianship / curatorship
* Patient under AME (state medical aid)

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Paediatric and adult patient treated by CAR-T cells
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-04-17 (Estimated); Study Completion 2025-04-17 (Estimated)

PRIMARY OUTCOMES:
Rate of CMV reactivation | Up to 3 months after inclusion
  Rate of CMV reactivation occurring within the first 3 months after CAR-T-cell infusion in paediatric and adult patients treated for refractory B cell acute lymphoblastic leukemia (B-ALL) and diffuse large B-cell lymphoma (DLBCL).

SECONDARY OUTCOMES:
Rate of CMV disease | Up to 3 months
Rate of anellovirus infection | Up to 3 months
Rate of pegivirus infection | Up to 3 months
Rate of redondovirus infection | Up to 3 months
Correlation between CMV reactivation and the occurrence of other bacterial or fungal infections | Up to 3 months
Correlation between CMV reactivation and the expansion of CAR-T cells | Up to 3 months
Correlation between CMV reactivation and other early viral persistent reactivations (anellovirus, pegivirus, redondovirus) | Up to 3 months
Rate of CMV reactivation in patients with acute leukemia | Up to 3 months
Rate of CMV reactivation in patients with lymphoma | Up to 3 months
Detection of mutations in the CMV DNA polymerase gene in patients under acyclovir or valacyclovir prophylaxis | Up to 3 months
Health related quality of life (HRQL)) of the study population with or without CMV activation | Up to 3 months
  EQ-5D-5L scale (adult) EQ-5D-Y scale (child) First part describes 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) Second part is a visual analogue scale with a score varying from 0 to 100; the higher the score the better the state of health.
Cost of illness of CMV disease | Up to 3 months
  Illness of CMV disease is defined by prolonged initial hospitalization, additional hospitalizations, increased surveillance in case of reactivation (consults and biological sampling), treatments)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hopital Robert Debré - APHP, Paris
  - Hopital Saint Louis - APHP - Service d'hématologie " Unité Adolescents et jeunes adultes ", Paris
  - Hopital Saint-Louis - APHP - Service d'éhamotologie - oncologie, Paris

IPD SHARING:
Plan to Share IPD: Undecided